CLINICAL TRIAL: NCT04604483
Title: Percutaneous Tibial Nerve Stimulation for Chronic Anal Fissure - a Prospective Study
Brief Title: Percutaneous Tibial Nerve Stimulation (PTNS) for the Treatment of Chronic Anal Fissure
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTNS for anal fissure
Record Dates: First submitted 2020-10-14; First posted 2020-10-27 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Fissure in Ano
Keywords: Anal fissure; Percutaneous Tibial Nerve Stimulation; PTNS
MeSH Terms: conditions — Fissure in Ano

STUDY DESIGN:
Intervention Model Description: Prospective non-randomized trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PTNS (Experimental): Treatment with PTNS for chronic anal fissure, treatment to be given for 30 minutes during 10 consecutive work Days.
  Interventions: Device: PTNS

INTERVENTIONS:
Device: PTNS — Patients meeting the criteria are treated with PTNS and are evaluated at 3 months and 1 year after end of treatment.
  Other Names: Percutaneous Tibial Nerve Stimulation

SUMMARY:
Chronic anal fissure rarely heals spontaneously. About 50% heal on administration om topical muscle relaxants (e.g. diltiazem) and/or injection of Botulinum toxin, but for the remainder of patients surgery (with lateral internal sphincterotomy or fissurectomy) with subsequent risks of anal incontinence has been the golden standard. Treatment with PTNS (percutaneous tibial nerve stimulation) has been showed to produce healing of chronic anal fissures not responding to topical treatment, thus avoiding the risk for debilitating anal incontinence.

DETAILED DESCRIPTION:
This study will prospectively include 52 patients with chronic anal fissure that have received topical treatment and stool softeners and have all been evaluated by experienced proctological surgeons. The treatment will be given for 10 consecutive work days and then evaluated at 3 and 12 months. If the patients symptoms are unimproved at 3 months alternative treatments will be offered.

ELIGIBILITY:
Inclusion Criteria:

* Verified anal fissure (Clinical assessement by experienced proctological surgeon)
* Full conservative treatment has been given

Exclusion Criteria:

* Inflammatory bowel disease
* Fistula and/or anal abscess
* Patients with compromised immunity
* Pregnancy
* Treatment with anti-coagulants (not aspirin)
* Previous irradiation towards pelvic floor
* Pacemaker or implanted defibrillator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Healing rate | 3 months after treatment
  Healing of anal fissure from assessement of clinical and/or data from patient form
Healing rate | 12 months after treatment
  Healing of anal fissure from assessement of clinical and/or data from patient form

SECONDARY OUTCOMES:
Bowel movements | 3 months after treatment
  Changes in frequency of bowel emptying and consistency of bowel contents Before and after treatment
Bowel movements | 12 months after treatment
  Changes in frequency of bowel emptying and consistency of bowel contents Before and after treatment
Adverse effects | 3 months after treatment
  Reports of adverse effects (subjective/objective)
Adverse effects | 12 months after treatment
  Reports of adverse effects (subjective/objective)
Smoking | 3 months after treatment
  Differences in healing rates between smokers and non-smokers
Smoking | 12 months after treatment
  Differences in healing rates between smokers and non-smokers

CONTACTS AND LOCATIONS:
Overall Officials: Louis B Johnson, PhD, Principal Investigator — Lund University
Locations (1):
- Skåne University Hospital, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: No
No intention to make individual participant data available to other researchers

REFERENCES:
- [Background] Nelson RL, Thomas K, Morgan J, Jones A. Non surgical therapy for anal fissure. Cochrane Database Syst Rev. 2012 Feb 15;2012(2):CD003431. doi: 10.1002/14651858.CD003431.pub3. PMID 22336789